CLINICAL TRIAL: NCT03277573
Title: A Phase 1b, 12-Month, Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of Salsalate in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Salsalate in Patients Mild to Moderate Alzheimer's Disease
Acronym: SAL-AD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adam Boxer (Other)
Responsible Party: Sponsor-Investigator, Adam Boxer, Director, Alzheimer's Disease and Frontotemporal Dementia Clinical Trials Program, Professor of Neurology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UC-SAL-AD-001
Record Dates: First submitted 2017-07-27; First posted 2017-09-11 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
Keywords: Salsalate
MeSH Terms: conditions — Alzheimer Disease | interventions — salicylsalicylic acid

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind study. Only investigational pharmacist will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Salsalate (Experimental): Drug: Salsalate 2 tablets twice daily (3,000 mg total daily) by mouth for 12 months
  Interventions: Drug: Salsalate
- Placebo (Placebo Comparator): Drug: Placebo 2 tablets twice daily by mouth for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salsalate — Salsalate is a non-acetylated dimer of salicylic acid, and is classified as a non-steroidal anti-inflammatory drug (NSAID). Salsalate has been commercially available in the US as a prescription drug for the relief of the signs and symptoms of rheumatoid arthritis, osteoarthritis, and related rheumatic disorder for decades.
  Arms: Salsalate
Drug: Placebo — Inactive ingredient
  Arms: Placebo

SUMMARY:
The purpose of the study is to test the safety and tolerability of twice daily Salsalate in patients with mild to moderate Alzheimer's Disease. Half of the participants will receive Salsalate and half will receive placebo during the 1-year duration of the study.

DETAILED DESCRIPTION:
This is a Phase 1b, 12-month, randomized, double-blind, placebo-controlled study of the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of salsalate in patients with mild to moderate AD. Approximately 40 subjects will be randomized 1:1 to placebo or active. All study drugs will be administered orally bid [two placebo tablets bid or two 750 mg salsalate tablets bid (for a total daily dose of 3,000 mg)] for 12 months.

This study will test the effects of Salsalate on cerebrospinal fluid (CSF) proteins, brain magnetic resonance imaging (MRI), and cognitive (thinking and memory) tests in subjects with mild to moderate AD. This study uses placebo which looks like the experimental drug but does not have any active drug in it.

ELIGIBILITY:
Inclusion Criteria:

1. Between 50 and 85 years of age (inclusive);
2. Meets National Institute on Aging-Alzheimer's Association Workgroups criteria for probable AD dementia (McKhann et al. 2011) (30);
3. MRI at Screening is consistent with AD (≤ 4 microhemorrhages, and no large strokes or severe white matter disease);
4. MHIS at Screening is ≤ 4;
5. MMSE at Screening is between 14 and 30 (inclusive);
6. FDA-approved AD medications are allowed as long as the dose is stable for 2 months prior to initial Screening visit. Other medications (except those listed under exclusion criteria) are allowed as long as the dose is stable for 30 days prior to initial Screening visit;
7. Has a reliable study partner who agrees to accompany the subject to visits, and spends at least 5 hours per week with the subject;
8. Agrees to the lumbar puncture and CSF collection at Screening and after 11.5 months of study drug administration. The lumbar puncture and CSF collection at the end of Month 6 is optional and is not required for eligibility;
9. Positive amyloid PET scan at Screening. Previous amyloid PET scan positivity or previous AD biomarker (Aβ/tau level) positivity may be used instead of performing an amyloid PET scan at Screening at the Investigator's discretion;
10. Signed and dated written informed consent obtained from the subject and the subject's caregiver in accordance with local IRB regulations;
11. Males and all WCBP agree to abstain from sex or use an adequate method of contraception for the duration of the study and for 30 days after the last dose of study drug.

Exclusion Criteria:

1. Any medical condition other than AD that could account for cognitive deficits (e.g., active seizure disorder, stroke, vascular dementia);
2. History of negative AD biomarker studies (CSF Aβ/tau levels or amyloid PET), or a negative amyloid PET scan during Screening;
3. History of significant cardiovascular, hematologic, renal, or hepatic disease (or laboratory evidence thereof);
4. Systolic blood pressure exceeding 180 mmHg or diastolic blood pressure exceeding 100 mmHg at Screening or Baseline;
5. History of peptic ulcer disease or GI bleeding;
6. History of asthma, urticaria, or allergic-type reactions after taking NSAIDs or aspirin;
7. History of aspirin triad (i.e., aspirin allergy, nasal polyps, and asthma);
8. History of autoimmune disorders deemed clinically significant by the Investigator;
9. History of major psychiatric illness or major depression that in the opinion of the Investigator would pose a safety risk or interfere with the appropriate interpretation of study data;
10. Neutrophil count <1,500/mm3, platelets <100,000/mm3, serum creatinine >1.5 x upper limit of normal (ULN), total bilirubin >1.5 x ULN, alanine aminotransferase (ALT) >3 x ULN, aspartate aminotransferase (AST) >3 x ULN, or INR >1.2 at Screening;
11. Evidence of any clinically significant findings on Screening or baseline evaluations which, in the opinion of the Investigator would pose a safety risk or interfere with appropriate interpretation of study data;
12. Current or recent history (within four weeks prior to Screening) of a clinically significant bacterial, fungal, or mycobacterial infection;
13. Current clinically significant viral infection. Subjects with chicken pox, influenza, or flu symptoms are not eligible;
14. Major surgery within four weeks prior to initial Screening visit;
15. Unable to tolerate MRI scan at Screening;
16. Any contraindication to or unable to tolerate lumbar puncture at Screening, including use of anti-coagulant medications such as warfarin. Daily administration of 81 mg aspirin will be allowed as long as the dose is stable for 30 days prior to initial Screening visit;
17. Chronic use of other NSAIDs or salicylates for any reason, except for daily baby aspirin (81 mg);
18. Chronic use of oral corticosteroids or other immunosuppressants;
19. Subjects who, in the opinion of the Investigator, are unable or unlikely to comply with the dosing schedule or study evaluations;
20. Participation in another AD clinical trial within 3 months of initial Screening visit or treatment with another investigational drug within 30 days of initial Screening visit;
21. Known hypersensitivity to the inactive ingredients in the study drug (placebo or active);
22. Pregnant or lactating;
23. Positive pregnancy test at Screening or Baseline (Day 1);
24. Cancer within 5 years of initial Screening visit, except for non-metastatic skin cancer or prostate cancer without signs of metastasis

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 months
  Assess adverse events during 12 months administration of Salsalate or Placebo

SECONDARY OUTCOMES:
Changes in Pharmacokinetic properties of Salsalate in Plasma and Cerebrospinal Fluid | 6; 11.5 months
  Measure steady-state plasma and cerebrosinal fluid concentrations of salsalate and its metabolites.
Changes in Pharmacodynamic properties of Salsalate in Cerebrospinal Fluid | 6; 11.5 months
  Measure CSF concentrations of total tau, phosphorylated tau, and neurofilament light chain

OTHER OUTCOMES:
Change in brain volume on brain MRI | 6; 12 months
  Measure of global and regional volumes of interest (such as hippocampus)
Change in structural and functional connectivity on brain MRI | 6; 12 months
  Connectivity between brain regions measured using diffusion tensor MRI and resting state functional MRI
Change in Cerebrospinal Fluid Biomarkers of phosphorylated tau | 6; 11.5 months
  Measure CSF concentrations of phosphorylated tau protein (p-tau) pg/mL
Change in Cerebrospinal Fluid Biomarkers of neurofilament light chain | 6; 11.5 months
  Measure CSF concentrations of neurofilament light chain protein (NfL) pg/ml
Change in Cerebrospinal Fluid Biomarkers of total tau | 6; 11.5 months
  Measure CSF concentrations of total tau protein (t-tau) pg/mL
Change in Cerebrospinal Fluid Biomarkers of beta amyloid 1-42 | 6; 11.5 months
  Measure CSF concentrations of beta amyloid protein (Abeta1-42) pg/mL
Change in Alzheimer's Disease Assessment Scale-cognitive scale | 6;12 months
  Measure changes using the Alzheimer's Disease Assessment Scale-cognitive (ADAS-cog) which evaluates cognitive dysfunctions
Change in Mini Mental State Examination | 6;12 months
  Measure changes using the Mini Mental State Exam (MMSE) which evaluates cognitive function.
Change in Alzheimer's disease Clinical Activities of Daily Living Scale | 6;12 months
  Measure changes in function, and in particular the degree of disability using the Alzheimer's disease Clinical Activities of Daily Living scale (ADCS-ADL)
Change in Clinical Dementia Rating Scale (CDR-SB) | 6;12 months
  Measure change in dementia status using the Clinical Dementia Rating scale (CDR-SB)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Boxer, MD, PhD, Principal Investigator — UCSF Memory and Aging Center
Locations (2):
- United States (2):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Min SW, Chen X, Tracy TE, Li Y, Zhou Y, Wang C, Shirakawa K, Minami SS, Defensor E, Mok SA, Sohn PD, Schilling B, Cong X, Ellerby L, Gibson BW, Johnson J, Krogan N, Shamloo M, Gestwicki J, Masliah E, Verdin E, Gan L. Critical role of acetylation in tau-mediated neurodegeneration and cognitive deficits. Nat Med. 2015 Oct;21(10):1154-62. doi: 10.1038/nm.3951. Epub 2015 Sep 21. PMID 26390242
- [Background] Montine TJ, Larson EB. Late-life dementias: does this unyielding global challenge require a broader view? JAMA. 2009 Dec 16;302(23):2593-4. doi: 10.1001/jama.2009.1863. No abstract available. PMID 20009062
- [Background] Jack CR Jr, Holtzman DM. Biomarker modeling of Alzheimer's disease. Neuron. 2013 Dec 18;80(6):1347-58. doi: 10.1016/j.neuron.2013.12.003. PMID 24360540
- [Background] Green RC, Schneider LS, Amato DA, Beelen AP, Wilcock G, Swabb EA, Zavitz KH; Tarenflurbil Phase 3 Study Group. Effect of tarenflurbil on cognitive decline and activities of daily living in patients with mild Alzheimer disease: a randomized controlled trial. JAMA. 2009 Dec 16;302(23):2557-64. doi: 10.1001/jama.2009.1866. PMID 20009055
- [Background] Gauthier S, Aisen PS, Ferris SH, Saumier D, Duong A, Haine D, Garceau D, Suhy J, Oh J, Lau W, Sampalis J. Effect of tramiprosate in patients with mild-to-moderate Alzheimer's disease: exploratory analyses of the MRI sub-group of the Alphase study. J Nutr Health Aging. 2009 Jun;13(6):550-7. doi: 10.1007/s12603-009-0106-x. PMID 19536424
- [Background] Holmes C, Boche D, Wilkinson D, Yadegarfar G, Hopkins V, Bayer A, Jones RW, Bullock R, Love S, Neal JW, Zotova E, Nicoll JA. Long-term effects of Abeta42 immunisation in Alzheimer's disease: follow-up of a randomised, placebo-controlled phase I trial. Lancet. 2008 Jul 19;372(9634):216-23. doi: 10.1016/S0140-6736(08)61075-2. PMID 18640458
- [Background] Doody RS, Thomas RG, Farlow M, Iwatsubo T, Vellas B, Joffe S, Kieburtz K, Raman R, Sun X, Aisen PS, Siemers E, Liu-Seifert H, Mohs R; Alzheimer's Disease Cooperative Study Steering Committee; Solanezumab Study Group. Phase 3 trials of solanezumab for mild-to-moderate Alzheimer's disease. N Engl J Med. 2014 Jan 23;370(4):311-21. doi: 10.1056/NEJMoa1312889. PMID 24450890
- [Background] Salloway S, Sperling R, Fox NC, Blennow K, Klunk W, Raskind M, Sabbagh M, Honig LS, Porsteinsson AP, Ferris S, Reichert M, Ketter N, Nejadnik B, Guenzler V, Miloslavsky M, Wang D, Lu Y, Lull J, Tudor IC, Liu E, Grundman M, Yuen E, Black R, Brashear HR; Bapineuzumab 301 and 302 Clinical Trial Investigators. Two phase 3 trials of bapineuzumab in mild-to-moderate Alzheimer's disease. N Engl J Med. 2014 Jan 23;370(4):322-33. doi: 10.1056/NEJMoa1304839. PMID 24450891
- [Background] Luna-Medina R, Cortes-Canteli M, Sanchez-Galiano S, Morales-Garcia JA, Martinez A, Santos A, Perez-Castillo A. NP031112, a thiadiazolidinone compound, prevents inflammation and neurodegeneration under excitotoxic conditions: potential therapeutic role in brain disorders. J Neurosci. 2007 May 23;27(21):5766-76. doi: 10.1523/JNEUROSCI.1004-07.2007. PMID 17522320